CLINICAL TRIAL: NCT04024124
Title: CART Phase 3 Study: Diagnostic Performance of a Ring-type Wearable Device Using Deep Learning Analysis of Photoplethysmographic Signals for Detecting Atrial Fibrillation Among Ambulatory Patients
Brief Title: A Ring-type Wearable Device for Atrial Fibrillation Among Ambulatory Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Sky Labs Inc. (Unknown)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Other Study IDs: CART3
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Deep learning; Diagnosis; Photoplethysmography; Wearable electronic devices
MeSH Terms: conditions — Atrial Fibrillation; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates diagnostic performance of a ring-type wearable device for detecting atrial fibrillation. This is a prospective cohort registry study began after the date of IRB approval and until 31th Dec. 2023. The eligible criteria are (1) those who admitted the institution for elective direct-current cardioversion or catheter ablation of persistent atrial fibrillation, (2) those who were successfully converted to sinus rhythm after the intervention, and (3) aged 19 years or more. The exclusion criteria are (1) those aged less than 19 years, (2) those who are not converted to sinus rhythm after the intervention, and (3) those who are not eligible to measure photoplethysmographic signals. This study aims to recruit 100 participants in total. The participants are required to record photoplethysmographic signals by the ring device in addition to routine procedures of direct-current cardioversion or catheter ablation, hence, the study is at minimal risk.

DETAILED DESCRIPTION:
1. Study title: Diagnostic Performance of a Ring-type Wearable Device Using Deep Learning Analysis of Photoplethysmographic Signals for Detecting Atrial Fibrillation Among Ambulatory Patients.
2. Study type: Investigator initiated study.
3. Study design: Prospective observational cohort registry design.
4. Sponsor: Sky Labs, Inc., Republic of Korea.
5. The aim of the study: To evaluate diagnostic performance of a ring-type wearable device for detecting atrial fibrillation among ambulatory patients.
6. Study period: From the date of IRB approval to 31th Dec. 2023.
7. The size of study population: 100 participants
8. The eligibility criteria:

(1) Those with persistent atrial fibrillation (2) Those who admitted the institution for elective direct-current cardioversion or catheter ablation (3) Those who are successfully converted to sinus rhythm (4) Those aged 19 years or more

9. The exclusion criteria:

1. Those with other forms of cardiac arrhythmias
2. Those aged less than 19 years
3. Those who are not eligible to perform electrical cardioversion or catheter ablation
4. Those who are not converted to sinus rhythm after the intervention

10. Procedures of the study

1. A participant is under the routine procedures of direct- current cardioversion or catheter ablation.
2. On admission, a participant is given with detailed information of the study.
3. After the informed consent, the only additional procedure due to the study is recording photoplethysmographic signal by wearing a ring-type device. The participant is instructed how to use the ring device.
4. Recorded signals are evaluated without encompassing persornal information.
5. The participant is required to wear the ring device and Holter monitoring device, and record his or her photoplethysmographic signals with ambulatory electrocardiography during the day. The ring is designed to automatically record user's photoplethysmographic signals and wirelessly transmit the data to user's smartphone. Detailed timings of wearing on/off the ring device and the Holter device are informed by a designated research crew.
6. The participant visits outpatient clinic as scheduled accordingly. At the clinic, the participant returns the ring device, Holter monitoring device, and the recorded data to the designated researcher crew.
7. Throughout the study, there is no intervention to the participants. The only additional step due to the participation of the study is that wearing the ring device and Holter monitoring device during their daily lives until the next outpatient clinic.

11. Financial benefits to the participants: None.

ELIGIBILITY:
Inclusion Criteria:

* Those with persistent atrial fibrillation
* Those who admitted for elective direct-current cardioversion or catheter ablation
* Those who are successfully converted to sinus rhythm
* Those who aged 19 years or more

Exclusion Criteria:

* Those who aged less than 19 years
* Those who had other types of cardiac arrhythmias
* Those who are not eligible to perform electrical cardioversion or catheter ablation
* Those who are not converted to sinus rhythm

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study consecutively recruits participants who admitted for elective direct-current cardioversion or catheter ablation due to persistent atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | 1 month (from the discharge to the next outpatient clinic)
  Diagnostic performance of a ring-type wearable device for detecting atrial fibrillation (parameters including sensitivity, specificity, positive predictive value, negative predictive value).

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, MD, PhD, Principal Investigator — Devision of Cardiology, Department of Internal Medicine, Seoul National University Hospital
Locations (1):
- Seoul National university Hostpital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Currently, according to the decision with IRB of the institution, the IPD is not planned to be shared with other researchers for the purpose of protecting potential privacy issues of the participants.